CLINICAL TRIAL: NCT05633420
Title: A Multi-Center Single Arm, Open-label, Pilot Clinical Trial to Explore Efficacy and Safety of Pyramax in Mild to Moderate COVID-19 Patients
Brief Title: Pilot Clinical Trial to Explore Efficacy and Safety of Pyramax in Mild to Moderate COVID-19 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-PA-COV-204
Record Dates: First submitted 2022-11-30; First posted 2022-12-01 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: Pyramax; pyronaridine-artesunate; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyramax (Experimental): pyronaridine-artesunate (180/160 mg)
  Interventions: Drug: Pyramax

INTERVENTIONS:
Drug: Pyramax — Participant body weight
  * ≥65 kg (Pyramax 4 tablets)
  * ≥45 kg and <65 kg (Pyramax 3 tablets)
  Other Names: pyronaridine-artesunate

SUMMARY:
This study is a multi-center, single-arm, open-label, pilot clinical trial to explore efficacy and safety of Pyramax in mild to moderate COVID-19 patients

DETAILED DESCRIPTION:
This study is a multi-center, single-arm, open-label, pilot clinical trial to explore the efficacy and safety of Pyramax Tab. in patients diagnosed with mild to moderate Coronavirus Disease-19 (COVID-19).

Major inclusion criteria are eligible patients confirmed with mild or moderate COVID-19, along with one or more symptoms in association with COVID-19 within 5 days (120 hours) before the screening, who do not need adjunctive oxygen therapy.

Subjects eligible to participate in this study will be enrolled and will take Investigational Product once a day for 3 days.

Subjects will participate in this study for 29 days in total, and subjects will follow the procedure in accordance with the Schedule of Clinical Trial Events to evaluate efficacy and safety after administration of Investigational Product.

Even though subjects are released from quarantine or discharged after showing clinical improvements, subjects should continue to visit hospitals for follow-up until 29 days in accordance with scheduled visit. The criteria of specific discharge (release from quarantine) for confirmed COVID-19 patients with symptoms should follow the latest version of the infectious disease prevention and control guideline.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Patients with body weight ≥45 kg at screening
* Patients who were first confirmed with COVID-19 through Real-Time Polymerase Chain Reaction (RT-PCR) or antigen test within 96 hours of baseline (those who have no history of confirmed COVID-19 within 3 months from the time of screening)
* Patients confirmed with mild or moderate COVID-19, along with one or more symptoms in association with COVID-19 within 5 days (120 hours) before screening, who do not need adjunctive oxygen therapy
* Patients who are fully informed of this study, voluntarily decide to participate in this study and provide written consent to comply with requirements for this study

Exclusion Criteria:

* Patients with severe or critical COVID-19
* Patients requiring hospitalization for therapeutic purposes for COVID-19 such as oxygen therapy or higher level of care, or who may be potentially transferred to another hospital other than the institution within 72 hours, with decreased oxygen saturation (<94%) at screening.
* Patients who have received or who have plans to receive any anti-viral drugs to treat COVID-19 infection or medications that may affect the course of treatment within 28 days before participating in this study or before a sufficient wash-out period
* Patients with a known allergic reaction to the active ingredients (pyronaridine tetraphosphate, artesunate) and other ingredients of investigational product
* Patients with a gastrointestinal disease or who underwent a surgery that can affect the absorption, distribution, metabolism and excretion of the drug, or who have active gastritis, gastrointestinal tract/rectal bleeding, gastric ulcer, and pancreatitis or pancreatic function abnormalities (excluding general appendectomy or hernia repair surgery)
* Patients who cannot be orally administered investigational product
* Pregnant, breast-feeding or females with positive pregnancy test at screening
* Females and males who have a child-bearing plan or who are unwilling to commit to the use of the highly effective methods of contraception during the study period and for 3 months after the study period, such as combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, sexual abstinence and surgical sterilization (vasectomy, tubal ligation, etc.)
* Patients whom the investigator considers inappropriate for the study due to chronic underlying disease or other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-24 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Time to negative conversion of COVID-19 infectious viable virus after administration of the investigational product | follow up to Day29
  Time took for subjects with positive infectious viable virus from virus culture at the baseline to get first negative infectious virus test result

SECONDARY OUTCOMES:
Change from baseline in SARS-CoV-2 infectious virus titer by viral culture | follow up to Day14
  Changes in COVID-19 infectious viral titer compared to the baseline
Change from baseline in SARS-CoV-2 RNA load by quantitative RT-PCR | follow up to Day14
  Changes in COVID-19 viral RNA load compared to the baseline
Percentage of subjects requiring acute treatment for more than 24 hours in a hospital or acute treatment facility due to COVID-19 or who have died until 29 days after administration | follow up to Day29
  Proportion of participants with progression to severe COVID-19 through Day 29 assessed by the composite outcome of COVID-19-related adjudicated hospitalization or oxygen therapy or more extensive care or death from any cause
Percentage of patients with new and aggravated pneumonia until 29 days after administration of the investigational product | follow up to Day29
  Defined as new occurrence or aggravation of existing pneumonia

OTHER OUTCOMES:
Time to sustained symptom resolution (score of 0 to 1) on 11-point World Health Organization Clinical Progression Scale after administration of the investigational product | follow up to Day29
  Time to sustained symptom resolution [defined as the instance of the first asymptomatic status (score of 0 to 1) for ≥96 hours on the 11-point World Health Organization Clinical Progression Scale for clinical symptoms]
Time to sustained symptom resolution of all COVID-19-related symptoms for ≥96 hours | follow up to Day29
  Defined symptoms include congestion or runny nose, sore throat, cough, fever, fatigue, shortness of breath or difficulty breathing, chills, muscle or body aches, headache, nausea, vomiting, diarrhea, loss of smell, loss of taste and other symptoms associated with COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Yee Gyung Kwak, MD, Phd, Principal Investigator — Inje University Ilsan Paik Hospital; Jin Soo Lee, MD, Phd, Principal Investigator — Inha University Hospital
Locations (2):
- South Korea (2):
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Inha University Hospital, Incheon

IPD SHARING:
Plan to Share IPD: No